CLINICAL TRIAL: NCT05446363
Title: Glaucoma Telemedicine Screening
Acronym: GOLDING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Olomouc (Other)
Collaborators: Palacky University (Other)
Responsible Party: Principal Investigator, Ladislav Stanke, Principal Investigator, University Hospital Olomouc
Other Study IDs: GOLDING
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Medimonitor — A digital solution consisting of web based portal gathering data from mobile fundus camera and intraocular tonometer provided to the physicians located remotely to the University hospital that provides consults and analyses of on-site gathered data.

SUMMARY:
The incidence of glaucoma is currently growing in the world's population, including the younger ones. However, the number of specialists who could perform examinations is unavailable in many areas of the Czech Republic outside large agglomerations. There is suitable alternative procedure that would make it possible to increase the intensity of screening, for example in general practitioners surgeries via application of teleophthalmology. Early detection is absolutely essential for the patient (and therefore the health care system) for his/her further successful treatment. At the same time, all the necessary technical prerequisites are well known and commercially available.

DETAILED DESCRIPTION:
Detailed Description: The aim of this study is to increase the detection of patients suspected of having glaucoma. For this purpose, the use of a combination of a mobile fundus camera and a mobile intraocular tonometer is proposed. These devices are used within the general practitioners' surgeries in the rural parts of Olomouc and Jeseniky region. Their combination will allow a better stratification of patients suspected of glaucoma into the following groups:

* patients with ocular hypertension (higher intraocular pressure and normal optic disc)
* patients with normotensive glaucoma (normal intraocular pressure and suspected optic disc)
* glaucoma patients (higher intraocular pressure and suspected optic disc)

The advantage of involving a fundus camera is also in the possibility of the retinal pathologies detection such as diabetic retinopathy or age-related macular degeneration as a secondary outcome of the study.

However, the primary goal of the study is to detect glaucoma and ocular hypertension. This area is also supported by the Risk Factors Questionnaire and the Patient Education Questionnaire.

All patients will be evaluated by University hospital Olomouc (FNOL) ophthalmology specialists who will evaluate data coming through the specifically designed FNOL telemedicine webportal from intraocular tonometers and fundus cameras. Suspected patients will be invited to the FNOL Eye Clinic for follow-up assessment using other modalities - perimeter, OCT, stationary fundus camera, etc.

The secondary goal of the project is to create a database combining retinal images with intraocular pressure values, and data from other modalities in suspected patients who come to the FNOL for follow-up examinations. This goal will support the epidemiological study as well as it opens up the possibility of building a neural network over the database for easier classification of glaucoma patients in the future.

As cognitive impairments (for instance Alzheimer's disease) can also be inferred with the above-described equipment, patients are also presented with a questionnaire to examine their cognitive performance. Data collected with use of questionnaires will be also part of the database. Consequently, presenting the tertiary outcome of the described study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Informed written and verbal consent

Exclusion Criteria:

• Absence of collaboration (informed consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General public of remote regions without available specialized ophthalmology deparments.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful fundus imaging of 90 % enrolled patients. | 3 month
  90% of captured fundus images are useful for subsequent diagnostics by the ophthalmologist located remotely.
Successful intraocular pressure measurement of 90 % enrolled patients. | 3 month
  90% of measured intraocular pressures are useful for subsequent diagnostics by the ophthalmologist located remotely.
Invitation of all suspected patients within 1 month timeframe after the diagnosis to the premises of University hospital Olomouc for aditional assessment. | 4 month
  Patients that were identified as suspected by the funduscopy and intraocular tonometry are subsequently invited for further assessment into the hospital.
Successful stratification of 90 % enrolled patients into groups with use of intraocular tonometer. | 4 month
  Differentiation of 90 % enrolled patients into the following groups:
  * patients with ocular hypertension (higher intraocular pressure)
  * patients with normotensive glaucoma (normal intraocular pressure)
  * glaucoma patients (higher intraocular pressure)
Successful stratification of 90 % enrolled patients into groups with use of fundus camera. | 4 month
  Differentiation of 90 % enrolled patients into the following groups:
  * patients with ocular hypertension (normal optic disc)
  * patients with normotensive glaucoma (suspected optic disc)
  * glaucoma patients (suspected optic disc)

CONTACTS AND LOCATIONS:
Locations (1):
- Ordinace Pospíšil, Postřelmov, Czechia